CLINICAL TRIAL: NCT07091474
Title: Little Movers: Promoting Motor Development in Early Childhood Through Educational and Therapeutic Interventions
Brief Title: Promoting Motor Development in Infants and Toddlers Through Education and Early Detection
Acronym: Little-Movers
Status: Not yet recruiting | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: Little movers
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Typical Development
Keywords: motor development; education; prevention; family; early age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Families and Early Childhood Educators: This cohort includes families of children aged 0-36 months and early childhood educators enrolled in structured educational workshops. The intervention consists of age-specific sessions tailored to three cohorts (0-12 months, 13-24 months, 25-36 months). Sessions provide education on motor milestones, the role of play, early stimulation techniques, and early warning signs of motor delays. Parents, caregivers, and educators participate in interactive discussions, practical activities, and resource sharing to enhance knowledge and support early motor development.
  Interventions: Behavioral: Educational Workshops for Parents and Early Educators
- Infants (0-36 months): This cohort includes infants aged 0-36 months who will undergo motor development assessments using validated tools, including the Standardized Infant Hand Assessment (s-HAI), Ages and Stages Questionnaire (ASQ-3), Hammersmith Infant Neurological Examination (HINE), and Infant Motor Profile (IMP). Assessments are scheduled annually for typically developing infants and monthly for those at risk or showing early signs of motor delays.
  Interventions: Other: Motor Development Assessment in Children 0-36 Months

INTERVENTIONS:
Behavioral: Educational Workshops for Parents and Early Educators — A structured series of age-specific educational workshops designed for parents, caregivers, and early childhood educators of children aged 0-36 months. The workshops are organized into three cohorts (0-12 months, 13-24 months, 25-36 months) and focus on typical motor milestones, active play, early stimulation strategies, and recognition of early warning signs of motor delays. Sessions include interactive activities, discussions, and distribution of educational resources. Pre- and post-workshop surveys and semi-structured interviews are conducted to evaluate changes in knowledge and attitudes.
  Groups: Families and Early Childhood Educators
Other: Motor Development Assessment in Children 0-36 Months — Comprehensive motor development assessments performed on infants aged 0-36 months using validated tools (Standardized Infant Hand Assessment [s-HAI], Hammersmith Infant Neurological Examination [HINE], Infant Motor Profile [IMP], and Ages and Stages Questionnaire [ASQ-3]). These evaluations aim to collect normative data on typical early motor development and to identify early signs of motor delays or neurological conditions, enabling timely referral and intervention. Assessments are conducted annually for typically developing infants and monthly for those identified as at risk.
  Groups: Infants (0-36 months)

SUMMARY:
The "Little Movers" study promotes healthy motor development in early childhood by providing education to caregivers and professionals in the child's environment and by implementing early detection strategies for motor delays.

The primary prevention component includes structured educational workshops designed for three age groups: 0-12 months, 13-24 months, and 25-36 months. These workshops focus on typical motor milestones, the importance of active play, early stimulation strategies, and how to recognize early warning signs of motor development delays. Participation impact will be measured using pre- and post-workshop surveys and semi-structured interviews with parents, caregivers, and educators.

The secondary and tertiary prevention component consists of a longitudinal observational study that follows infants aged 0 to 12 months. Motor development will be assessed using validated tools, including the Standardized Infant Hand Assessment (s-HAI), the Hammersmith Infant Neurological Examination (HINE), the Infant Motor Profile (IMP), and the Ages and Stages Questionnaire (ASQ-3). Infants with typical development will be reassessed annually, while those at risk or showing signs of motor delay will be monitored monthly. The goal is to detect motor delays as early as possible to allow timely referral and intervention.

ELIGIBILITY:
Inclusion Criteria (Workshops):

Legal guardians or primary caregivers of children aged 0 to 36 months enrolled in the participating daycare center. Early childhood educators working with children aged 0 to 36 months in the same center.

Inclusion Criteria (Observational Study):

Infants aged 0 to 12 months enrolled in the participating daycare center. Infants must not have a diagnosed neuromotor or neurological condition at the time of enrollment. Written informed consent must be obtained from a parent or legal guardian.

Exclusion Criteria:

Children with diagnosed neurological or genetic conditions affecting motor development. Families or educators who decline participation or do not provide informed consent. Children or families not enrolled in the participating daycare center.

Ages: 0 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population includes children aged 0 to 36 months with typical motor development who are enrolled in a participating kindergarten or early childhood education center. It also includes their primary caregivers (parents or legal guardians) and early childhood educators involved in the structured educational workshops.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver and educator knowledge and attitudes about motor development, as assessed with a 5-point Likert-scale questionnaire | Immediately before and immediately after each workshop session (same day)
  Knowledge and attitudes toward early motor development will be evaluated using a structured questionnaire administered immediately before and after workshop sessions. The questionnaire includes 10 items rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Total scores are calculated as the average of all items. Higher scores represent greater knowledge and more positive attitudes toward the importance of early motor milestones and play-based stimulation.
Neurological function in infants assessed by the Hammersmith Infant Neurological Examination (HINE) | Monthly assessments from 2 to 24 months of age.
  The Hammersmith Infant Neurological Examination (HINE) is a standardized clinical tool used to evaluate neurological function in infants aged 2 to 24 months. It includes domains such as cranial nerve function, posture, tone, and reflexes. The global score ranges from 0 to 78 points; higher scores indicate more typical neurological development. Scores below 40 in high-risk infants are associated with an increased probability of developing cerebral palsy.
Motor behavior in infants assessed by the Infant Motor Profile (IMP) | Monthly assessments from 3 to 18 months of age
  The Infant Motor Profile (IMP) is a standardized clinical assessment that evaluates the quality and variability of motor behavior in infants aged 3 to 18 months. The IMP provides scores across several domains (variation, adaptability, symmetry, fluency, and performance), with total scores calculated as a percentage (0-100%). Higher scores indicate more optimal and typical motor development. The assessment is designed to be repeated over time to monitor change in motor patterns, with results summarized as mean or change in percentage scores per assessment period.

SECONDARY OUTCOMES:
Unimanual hand function assessed by the Standardized Infant Hand Assessment (s-HAI) | Monthly from 3 to 12 months of age
  The s-HAI is a standardized tool to assess hand function in infants at risk for unilateral motor impairments. It evaluates spontaneous use of each hand during structured play activities. The total score ranges from 0 to 100 points. Higher scores reflect better unimanual hand performance. It is validated for use with infants between 3 and 12 months of age, particularly those with early signs of asymmetric movement or neurological risk factors.
Developmental progress assessed by Ages and Stages Questionnaire, Third Edition (ASQ-3) | Monthly from birth to 12 months of age
  The Ages and Stages Questionnaire, Third Edition (ASQ-3) is a parent-completed screening tool used to assess development in five domains: communication, gross motor, fine motor, problem solving, and personal-social skills, for children between 1 month and 5½ years. Each domain is scored separately, and results are compared to standardized age norms. Lower scores in any domain may indicate a risk of developmental delay. Scores are summarized for each domain and interpreted using established cut-off points.